CLINICAL TRIAL: NCT01465204
Title: Impact Evaluation of Large-Scale Sanitation and Hygiene Interventions in Peru, Tanzania, Senegal, Vietnam, Indonesia, and India
Brief Title: Impact Evaluation of Large-Scale Sanitation and Hygiene Interventions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Water and Sanitation Program, World Bank (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1095420
Record Dates: First submitted 2011-11-01; First posted 2011-11-04 (Estimated); Last update posted 2011-11-04 (Estimated); Status verified 2011-11

CONDITIONS: Infant Diarrhea
Keywords: Behavior Change; Hygiene & Sanitation Marketing
MeSH Terms: conditions — Diarrhea, Infantile

ARMS (4):
- Control (No Intervention)
- Handwashing Intervention (Experimental): scaling up handwashing with soap
  Interventions: Behavioral: Scaling Up Handwashing Behavior Change
- Sanitation Intervention (Experimental): total sanitation and sanitation marketing
  Interventions: Behavioral: Total Sanitation and Sanitation Marketing
- Combined (Experimental): combined scaling up handwashing with soap and total sanitation and sanitation marketing interventions
  Interventions: Behavioral: Total Sanitation and Sanitation Marketing; Behavioral: Scaling Up Handwashing Behavior Change

INTERVENTIONS:
Behavioral: Total Sanitation and Sanitation Marketing — Total Sanitation and Sanitation Marketing (TSSM) program is designed to promote demand for and supply of improved sanitation. On the demand side, it includes "Community-Led Total Sanitation" (CLTS). On the supply side, TSSM incorporates sanitation marketing interventions. Both CLTS and sanitation marketing draw heavily on the behavior-change communication and social marketing approaches that have been well developed in other sectors. The basic TSSM approach also builds sustainability and scalability through the strengthening of the national level sanitation sector enabling environment.
  Arms: Combined; Sanitation Intervention
Behavioral: Scaling Up Handwashing Behavior Change — The Handwashing with soap (HWWS) behavior change program expands and improves existing hygiene behavior change efforts with new and innovative promotional approaches in order to generate widespread and sustained improvement in handwashing with soap practices. These approaches include social marketing to deliver handwashing messages; broad and inclusive partnerships with government, private commercial marketing channels, and concerned consumer groups and NGOs.
  Arms: Combined; Handwashing Intervention

SUMMARY:
This study consists of an impact evaluation (IE) of the Scaling up Handwashing with Soap (HWWS) and Total Sanitation and Sanitation Marketing (TSSM) projects of the Water and Sanitation Program (WSP) of the World Bank. The objective of this study is to estimate the causal impact of the HWWS and TSSM interventions on the health and welfare of the rural poor in six developing countries: Peru, Tanzania, Senegal, Vietnam, Indonesia, and India. The IE will assess the impact of exposure to the HWWS and TSSM promotion on individual-level hygiene and sanitation practices, and on the health and welfare of children 0-5 years old. By introducing exogenous variation in handwashing and sanitation practices (through exposure to the HWWS and TSSM promotion), the IE will also answer a number of important questions related to the effect of the intended behavioral change (handwashing and improved sanitation) on health and welfare, thus providing information on the extent to which these behaviors alter intended development outcomes. This study uses a cluster-randomized experimental design, whereby the geographic units called clusters (e.g. village, commune, ward, depending on administrative structure of country) are randomly assigned to receive certain components of the Handwashing and Sanitation interventions in the case of treatment arms, and no Handwashing or Sanitation intervention in the case of control arms. . The final sample for the evaluation will consist of approximately 14,000 households, randomly selected, with at least one child between 0 and 24 months of age at baseline. Data will be collected from these 14,000 households (approximately 54,781 subjects) through household surveys, anthropometric measurements, blood and stool samples, direct observations of behaviors, and community surveys. The data collected will be analyzed using a differences in differences approach, where possible, and the results will be disseminated to country officials and others stakeholders.

ELIGIBILITY:
Inclusion Criteria:

* at least one child 0-24 months (at baseline) lives in the household
* adult family member (mother of primary caregiver of the selected children for the study) consents to participate in the study and provides consent for the child's participation

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 21878 (Actual)
Dates: Start 2007-11; Primary Completion 2010-12 (Actual); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Diarrhea in Children Under 5 | one year after the intervention
  incidence and prevalence of diarrhea and highly credible gastrointestinal illness (HCGI) in children under 5 years old (outcome measured in selected countries)

SECONDARY OUTCOMES:
ALRI in Children Under 5 | one year after the intervention
  incidence and prevalence of acute lower respiratory infections (ALRI) in children under 5 years old (outcome measured in selected countries)
Malnutrition in Children Under 5 | one year after the intervention
  prevalence of stunting, wasting and underweight in children under 5 years old by recording key anthropometric measurements (outcome measured in selected countries)
Anemia in Children Under 5 | one year after the intervention
  prevalence of anemia in children 6 months to 5 years old by measuring hemoglobin levels in the blood (outcome measured in selected countries)

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Gertler, PhD, Principal Investigator — UC Berkeley - Haas School of Business; Bertha Briceno, MPA/ID, Study Director — World Bank - Water and Sanitation Program; Alexandra Orsola-Vidal, MSc, Principal Investigator — World Bank - Water and Sanitation Program; Claire Chase, MSc, Principal Investigator — World Bank - Water and Sanitation Program; Sebastian F Galiani, PhD, Principal Investigator — Washington University School of Medicine; Sebastian W Martinez, PhD, Principal Investigator — Inter-American Development Bank; Paul M Wassenich, MPA, Principal Investigator — UC Berkeley; Alicia L Salvatore, MPH, PhD, Principal Investigator — Stanford University; Sumeet Patil, MA, Principal Investigator — Network for Engineering and Economics Research and Management; Manisha B Shah, PhD, Principal Investigator — UC Irvine; Lisa A Cameron, PhD, Principal Investigator — University of Melbourne; Jack M Colford, MD, MPH, PhD, Principal Investigator — UC Berkeley - School of Public Health; Ben Arnold, PhD, Principal Investigator — UC Berkeley; Lia CH Fernald, MBA, PhD, Principal Investigator — UC Berkeley - School of Public Health; Patricia K Kariger, PhD, Principal Investigator — UC Berkeley; Christine Stauber, PhD, Principal Investigator — Georgia State University - Institute of Public Health; Pavani K Ram, MD, Principal Investigator — University of Buffalo - SUNY

REFERENCES:
- [Derived] Briceno B, Coville A, Gertler P, Martinez S. Are there synergies from combining hygiene and sanitation promotion campaigns: Evidence from a large-scale cluster-randomized trial in rural Tanzania. PLoS One. 2017 Nov 1;12(11):e0186228. doi: 10.1371/journal.pone.0186228. eCollection 2017. PMID 29091726
- [Derived] Patil SR, Arnold BF, Salvatore AL, Briceno B, Ganguly S, Colford JM Jr, Gertler PJ. The effect of India's total sanitation campaign on defecation behaviors and child health in rural Madhya Pradesh: a cluster randomized controlled trial. PLoS Med. 2014 Aug 26;11(8):e1001709. doi: 10.1371/journal.pmed.1001709. eCollection 2014 Aug. PMID 25157929